CLINICAL TRIAL: NCT04465643
Title: Neoadjuvant Nivolumab Plus Ipilimumab for Newly Diagnosed Malignant Peripheral Nerve Sheath Tumor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Bristol-Myers Squibb (Industry); Congressionally Directed Medical Research Programs (U.S. Federal Agency); Cancer Research and Biostatistics Clinical Trials Consortium (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J20112; IRB00215437 (Other: Johns Hopkins University); W81XWH-22-1-0580 (Other: CDMRP Award Number)
Record Dates: First submitted 2020-07-07; First posted 2020-07-10 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Nerve Sheath Tumors
MeSH Terms: conditions — Nerve Sheath Neoplasms | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Immunotherapy with Nivolumab and Ipilimumab (Other): Nivolumab 4.5 mg/kg every 3 weeks (Q3W) x 2 Ipilimumab 1 mg/kg Q3W x 2 Nivolumab monotherapy 4.5mg/kg Q3W concurrent with standard therapy Nivolumab monotherapy should be held for at least 2 weeks before and 2 weeks after surgery
  Interventions: Drug: Nivolumab; Drug: Ipilimumab

INTERVENTIONS:
Drug: Nivolumab — Nivolumab 4.5 mg/kg Q3W x 2
Drug: Ipilimumab — Ipilimumab 1 mg/kg Q3W x 2

SUMMARY:
The purpose of the study is to evaluate safety and feasibility of neoadjuvant nivolumab plus ipilimumab prior to standard therapy (surgery, chemotherapy or radiation therapy) in patients with Neurofibromatosis Type 1 (NF1) and newly diagnosed pre-malignant and malignant peripheral nerve sheath tumors (MPNST) for whom surgery for resection of tumor is indicated.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of atypical neurofibromatous neoplasms of uncertain biologic potential (ANNUBP), low grade malignant peripheral nerve sheath tumor (MPNST) or high grade MPNST in accordance with the Miettinen et al diagnostic criteria via biopsy
* Plexiform neurofibroma or other tumors such as optic pathway glioma, other low-grade glioma or other neoplasm in addition to the ANNUBP, low grade MPNST or high grade MPNST that is stable (has not required treatment in the last 12 months and is not anticipated to need treatment in the next 12 months)
* Measureable disease by RECIST criteria in at least one site.
* Karnofsky Performance Scale ≥ 60%
* No contraindications for Nivolumab or Ipilimumab
* Normal organ and marrow function on routine laboratory tests
* Evidence of post-menopausal status or negative urinary/serum pregnancy test for female pre-menopausal subjects. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause
* Ability to understand and willingness of sign consent form
* Willingness to comply with the protocol for the duration of the study

Exclusion Criteria:

* Chemotherapy or other investigational agent for the current episode of newly diagnosed atypical neurofibroma or MPNST
* Prior therapy with an anti-PD-1, anti-PD-L1, or anti-PDL-2 antibody
* Known allergy to compounds of similar chemical or biologic composition to Nivolumab or Ipilimumab
* Pregnant or breastfeeding women
* Known history of Human Immunodeficiency Virus
* Active infection requiring therapy, including known positive tests for Hepatitis B surface antigen or Hepatitis C ribonucleic acid (RNA)
* Active autoimmune disease, history of autoimmune disease or history of syndrome that required systemic steroids or immunosuppressive medications, e.g. organ, tissue, or allogenic hematopoietic stem cell transplant (HSCT) recipients. Exceptions include those with resolved childhood asthma/atopy. Subjects with asthma who require intermittent use of bronchodilators (such as albuterol) will not be excluded from this study. Subjects are also permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger
* A condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
* Use of any vaccines against infectious diseases (e.g. varicella, influenza, etc.) up to 4 weeks (28 days) before receiving nivolumab and ipilimumab.
* Prisoners or subjects who are compulsorily detained for treatment of either a psychiatric or physical (e.g. infectious disease) illness
* Prior radiation doses equivalent to, or greater than, 8000 centigray (cGy) to the target lesions at 200 cGy fractions at any time point
* Any radiation to the the target lesions within 6 months of enrollment
* Other concurrent severe and/or uncontrolled medical disease, which could compromise participation in the study (e.g. uncontrolled diabetes, uncontrolled hypertension, severe infection, severe malnutrition, chronic liver or renal disease, active upper GI tract ulceration, congestive heart failure, etc.)

Ages: 12 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-06-08 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Safety of combination nivolumab and ipilimumab as assessed by number of participants who experience adverse events | Up to 2 years
  Number of participants who experience grade 1 or higher adverse events, as defined by Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v5.0).
Feasibility of combination nivolumab and ipilimumab as assessed by number of participants who experience adverse events | Up to 2 years
  Number of participants who experience grade 1 or higher adverse events, as defined by Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v5.0).
Maximum Tolerated Dose (MTD) as determined by number of participants with dose limiting toxicities (DLT) | Up to 2 years
  Maximum tolerated dose will be determined by the maximum dose at which the least number of participants experience dose-limiting toxicity. The dose limiting toxicity is defined using the Common Terminology Criteria for Adverse Events (CTCAE).
Feasibility of combination nivolumab and ipilimumab as assessed by number of participants who achieve a response | Up to 2 years
  Number of participants who achieve a response (improved progression free survival).

SECONDARY OUTCOMES:
Safety as assessed by number of treatment-emergent adverse events in patients on combination nivolumab and ipilimumab with NF1, standard low, or high grade MPNST therapy | Up to 2 years
  Number of participants who experience grade 1 or higher adverse events, as defined by Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v5.0)
Objective response rate (ORR) | Up to 2 years.
  Proportion of participants with measurable disease at baseline and have been re-evaluated after at least 1 cycle of therapy with observed reduction in tumor burden as defined by RECIST and iRECIST criteria after 2 doses of nivolumab and ipilimumab.
Change in pain levels in relation to target tumor as assessed by the Numeric Rating Scale | Baseline, Week 6, 4 months, and 8 months
  Evaluate pain levels in participants related to target tumor via the Numeric Rating Scale. Assessment to be performed at baseline, Week 6, 4 months, and 8 months via numeric grading scale (0 through 10) recorded by participant via survey in order to determine an improvement or worsening of pain throughout treatment. Lower scores indicate no pain or decreased levels of pain while higher score indicate increased levels of pain.
Change in pain levels in relation to target tumor as assessed by the Pain Interference Index | Baseline, Week 6, 4 months, and 8 months
  Evaluate pain in participants related to target tumor via the Pain Interference Index (6-24 years). Assessment to be performed at baseline, Week 6, 4 months, and 8 months via numeric grading scale (0 through 6) recorded by participant via survey In order to determine an improvement or worsening of pain throughout treatment. Lower scores indicate no interference or decreased levels of interference in every day life while higher scores indicate increased interference in ever day life.
Change in pain levels in relation to target tumor as assessed by the Patient-Reported Outcome Measurement Information System | Baseline, Week 6, 4 months, and 8 months
  Evaluate pain in participants related to target tumor via the Patient-Reported Outcome Measurement Information System (PROMIS). Assessment to be performed at at baseline, Week 6, 4 months, and 8 months via numeric grading scale (1 through 5) recorded by participant via survey in order to determine an improvement or worsening of pain throughout treatment. Higher scores indicate no to low difficulty in mobility while lower scores indicate increased difficulty or inability in mobility.

OTHER OUTCOMES:
Objective response rate (ORR) | At 4 months post intervention
  Proportion of participants who had measurable disease at baseline and have been re-evaluated after at least 1 cycle of therapy with observed reduction in tumor burden as defined by RECIST and iRECIST criteria at 4 months.
Progression Free Survival | Up to 2 years
  Proportion of participants who achieve progression free survival post treatment
Tumor Response as assessed by immune markers in tumor samples | Up to 2 years
  Analyses may include phosphorylated protines of signaling pathways and phenotypes of infiltrating immune cell populations including but not limited to CD3, CD4, FoxP3, CD25, CD8, CD45, CD11b, CD163, CD206, CD68, CD56, CD20, CD45RO and granzyme B. Pathologists will assign an intratumoral and peritumoral immune cell infiltrate grade of 0 through 3. Immunohistochemical analysis of exploratory markers will focus on areas including but not limited to: B7 family ligands PD-L1 (B7-H1), PD-L2 (B7-DC), B7-H3, B7-H4, as well as inhibitory receptors on lymphocytes, including PD-1, 2B4, LAG-3, BTLA, Tim-3, CTLA-4, and TIGIT.
Pharmacodynamic activity as assessed by markers in blood samples | Up to 2 years
  T cell subsets (including CD4, CD8, and Treg with CD25 and Foxp3) will be analyzed as well as co-stimulatory and co-inhibitory molecule expression and markers for T cell activation state (e.g., CD25, HLADR, CD45RO, LAP, PD-1, PD-L1, LAG-3, ICOS, OX40, 41BB). B cells (CD19, CD20, PD-1, PD-L1, PD-L2, ICOSL), dendritic cells and macrophages (CD68, CD83, CD1a, PD-L1, PD-L2, 4-1BB, 4-1BBL, ICOSL, HLA-DR) and natural killer cells (CD56) will be enumerated and characterized. Myeloid derived suppressor cells (MDSCs) will be enumerated by staining for CD14, CD11b, and HLADR expression.
CD3 Cell Count | Up to 1 year
  CD3 cell count in cells/mm^3
CD4 Cell Count | Up to 1 year
  CD4 cell count in cells/mm^3
FoxP3 Cell Count | Up to 1 year
  FoxP3 cell count in cells/mm^3
CD25 Cell Count | Up to 1 year
  CD25 cell count in cells/mm^3
CD8 Cell Count | Up to 1 year
  CD8 cell count in cells/mm^3
CD45 Cell Count | Up to 1 year
  CD45 cell count in cells/mm^3
CD11b Cell Count | Up to 1 year
  CD11b cell count in cells/mm^3
CD163 Cell Count | Up to 1 year
  CD163 cell count in cells/mm^3
CD206 Cell Count | Up to 1 year
  CD206 cell count in cells/mm^3
CD68 Cell Count | Up to 1 year
  CD68 cell count in cells/mm^3
CD56 Cell Count | Up to 1 year
  CD56 cell count in cells/mm^3
CD20 Cell Count | Up to 1 year
  CD20 cell count in cells/mm^3
CD45RO Cell Count | Up to 1 year
  CD45RO cell count in cells/mm^3
Granzyme B Cell Count | Up to 1 year
  Granzyme B cell count in cells/mm^3
PD-L1 Cell Count | Up to 1 year
  PD-L1 cell count in cells/mm^3
PD-L2 Cell Count | Up to 1 year
  PD-L2 cell count in cells/mm^3
B7-H3 Cell Count | Up to 1 year
  B7-H3 cell count in cells/mm^3
B7-H4 Cell Count | Up to 1 year
  B7-H4 cell count in cells/mm^3
PD-1 Cell Count | Up to 1 year
  PD-1 cell count in cells/mm^3
2B4 Cell Count | Up to 1 year
  2B4 cell count in cells/mm^3
LAG-3 Cell Count | Up to 1 year
  LAG-3 cell count in cells/mm^3
BTLA Cell Count | Up to 1 year
  BTLA cell count in cells/mm^3
Tim-3 Cell Count | Up to 1 year
  Tim-3 cell count in cells/mm^3
CTLA-4 Cell Count | Up to 1 year
  CTLA-4 cell count in cells/mm^3
TIGIT Cell Count | Up to 1 year
  TIGIT cell count in cells/mm^3
HLA-DR Cell Count | Up to 1 year
  HLA-DR cell count in cells/mm^3
LAP Cell Count | Up to 1 year
  LAP cell count in cells/mm^3
CD14 Cell Count | Up to 1 year
  CD14 cell count in cells/mm^3
ICOS Cell Count | Up to 1 year
  ICOS cell count in cells/mm^3
OX40 Cell Count | Up to 1 year
  OX40 cell count in cells/mm^3
4-1BB Cell Count | Up to 1 year
  4-1BB cell count in cells/mm^3
4-1BBL Cell Count | Up to 1 year
  4-1BBL cell count in cells/mm^3
ICOSL Cell Count | Up to 1 year
  ICOSL cell count in cells/mm^3
CD19 Cell Count | Up to 1 year
  CD19 cell count in cells/mm^3
CD1a Cell Count | Up to 1 year
  CD1a cell count in cells/mm^3

CONTACTS AND LOCATIONS:
Overall Officials: Jaishri Blakeley, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Medical Institution, Baltimore, Maryland, United States